CLINICAL TRIAL: NCT06313294
Title: Postoperative Follow-up Via Text Messages Automated Versus Telephone in Patients With Continuous Regional Anesthesia
Acronym: txt-RA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 230929002
Record Dates: First submitted 2024-02-23; First posted 2024-03-15 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Anesthesia; Regional Anesthesia; Nerve Pain
Keywords: Anesthesia, Regional; Regional Anesthesia; Continuous Nerve Block; Ambulatory; Outpatient follow-up
MeSH Terms: conditions — Neuralgia | interventions — Interviews as Topic

STUDY DESIGN:
Intervention Model Description: Participants will are assigned to one of two groups in parallel for the duration of the study
Who Masked: Participant
Masking Description: The research patients will be blind to the proposed intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App Group (Experimental): In this group the patients will use the app for asking about related to pain, patient satisfaction and another complications.
  Interventions: Other: Tracking application app
- Telephone interview group (Active Comparator): In this group the patients will receive the calling by one member of the healthcare team asking items related to pain, patient satisfaction and another complications.
  Interventions: Other: Telephone interview

INTERVENTIONS:
Other: Tracking application app — An app will be implemented for mobile monitoring in patients who use continuous postoperative ambulatory regional analgesia.
  Arms: App Group
Other: Telephone interview — Patients who use continuous postoperative outpatient regional analgesia will be followed up using the current traditional method of post-discharge telephone call.
  Arms: Telephone interview group

SUMMARY:
Monitoring performed by a trained operator has proven to be useful and valued by patients after the use of continuous regional anesthesia. A health professional calls each patient to gather information about their recovery. However, this direct communication strategy requires time and resources, especially if many patients are involved.

A modern and convenient approach involves the use of immediate communication technology for follow-up after a procedure. They may contain specific questions that patients can easily answer from their mobile devices.

Automated text messages could be associated with greater convenience and ease for patients with response rates at least like the traditional method. Phone calls, on the other hand, may be less scalable and require more human resources.

The objective of the project is to evaluate the feasibility of monitoring through automated electronic messaging by evaluating its usability using a validated scale in Spanish. response rate on the first day and adherence rate compared to that of the traditional method. Secondarily, adherence and differences in satisfaction will be compared.

DETAILED DESCRIPTION:
Communication with patients after performing any procedure under regional anesthesia is essential to evaluate pain control, measure patient satisfaction, and detect post-surgical and post-anesthetic complications.

However, for outpatients, achieving follow-up through phone calls can be a real challenge. Gessner et al report that successful daily telephone contact for patients discharged with a continuous perineural blocking catheter varies between 49 and 65%. While their results with the use of an automated messaging system, delivered results as promising as a response rate of 91%, considering a range of 18 to 90 years.

It is known that the mobile application market is expanding with great diversity on different devices. For this reason, there is great competition among application developers to create those that best fulfill the tasks proposed each day.

For this, the usability of mobile applications is a crucial tool to obtain a competitive advantage in these circumstances.

The significance of the expected results described above will open a door to the sequential or gradual implementation of a system that allows us to reduce the time and/or number of people required per day to achieve adequate follow-up of the patients. In addition, it would leave room for new projects that seek to devise an ordered work plan to identify the subgroup of patients who objectively require a live call to evaluate complications of the procedure.

The hypothesis is that the use of a mobile monitoring application in patients using postoperative continuous ambulatory regional analgesia is associated with usability levels equal to or higher than the 64th percentile measured on the SUS usability scale in its Spanish version.

To determine the degree of satisfaction that exists between the use of an automated system for the monitoring of patients undergoing continuous regional anesthesia at the UC-Christus Clinical Hospital. How much it impacts adherence to follow-up will also be reviewed, comparing it with the traditional method (telephone interview).

A convenience sample of 100 consecutive patients will be selected with continuous outpatient regional analgesia performed in the wards of the UC-Christus Clinical Hospital, San Carlos de Apoquindo Clinic and Santa Lucía Medical Center. For this, for a maximum period of 6 months, 100 patients will be randomly distributed into 2 groups, one for conventional telephone follow-up and the other for use of the app.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery with continuous ambulatory regional analgesia
* Able to understand, use and operate a smartphone to view the mobile application
* ASA I - II

Exclusion Criteria:

* Ages under 17 or over 76 years
* Emergency surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-05-31 (Actual); Primary Completion 2024-08-09 (Actual); Study Completion 2024-08-13 (Actual)

PRIMARY OUTCOMES:
Usability level of the tracking application | 1, 2 and 3 days after discharge.
  To determine the level of usability of the application using the SUS scale developed by John Brooke in 1986. This scale consists of 10 Likert-type statements. To calculate the result, the statements have an answer that will be equivalent to 1, 2, 3, 4 or 5, depending on said answer. The answers to the odd and even statements are added and then subtracted 5 and 25, respectively. The sum of both results is subsequently multiplied by 2.5 to obtain a result that ranges from 0 to 100, with 64 being our cut-off point to consider it acceptable.

SECONDARY OUTCOMES:
Patient satisfaction with Perception of Quality in Anesthesia | 1, 2 and 3 days after discharge.
  Measure and compare the level of patient satisfaction using the Perception of Quality in Anesthesia (PQA) scale validated in Spanish. In this instrument, the patient was asked to respond using a five-point Likert scale.
  The extremes of the scale were labelled 'very poor' to 'very good' or 'definitely not' to 'definitely yes' depending upon the question. Unsatisfactory patient responses were defined as a score of ≤3, any response 'yes' to the awareness question, or any description of nausea or vomiting in the PONV question.
  A quality index was calculated for each PQA question by multiplying the importance score against the performance score.
Patient adherence | 1, 2 and 3 days after discharge.
  Measure and compare patient adherence using the app versus the telephone follow-up method, defined as rate of response during the three days of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Altermatt, MD, Study Chair — Pontificia Universidad Catolica de Chile
Locations (1):
- Pontificia Universidad Catolica de Chile, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Derived] Strange E, Altermatt FR, Caceres L, Morrison C, Cortes L, Sumonte N, Neyem A; FAR-UC Group. Postoperative follow-up by automated text messaging versus telephone call in outpatient care with continuous regional analgesia: a randomized controlled feasibility trial. Reg Anesth Pain Med. 2025 Sep 18:rapm-2025-106818. doi: 10.1136/rapm-2025-106818. Online ahead of print. PMID 40973445